CLINICAL TRIAL: NCT02514057
Title: Gastrointestinal Symptom Questionnaire Validation
Status: Withdrawn | Type: Observational
Why Stopped: investigator emigrated
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Other Study IDs: 150725
Record Dates: First submitted 2015-07-31; First posted 2015-08-03 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Those With and Without Gastrointestinal Disorders
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy: Volunteers over 18 years
  Interventions: Other: Questionnaire
- Gastrointestinal disorders: Over 18 and with any gastrointestinal or liver disorder
  Interventions: Other: Questionnaire
- Non-gastrointestinal disorders: Over 18 and with any medical condition requiring hospital attention in which there is no primary gastrointestinal or liver disease
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Form filling only

SUMMARY:
Assessment of a new gastrointestinal symptom questionnaire in comparison to 2 well established and validated questionnaires that do not fully fit the requirements of an investigator concerned about gastrointestinal side effects in a patient without primary gastrointestinal disease.

DETAILED DESCRIPTION:
210 subjects Healthy (n=70), ill with non-GI disease (n=70), with GI disease (n=70) Age above 18 COnsent after full explanation Each subject completes 3 questionnaires Glasgow Dyspepsia Score Gastrointestinal Symptom Rating Scale New score This is a total of 48 questions Analysis will seek to validate the new score. There is no other intervention and no risks are anticipated.

ELIGIBILITY:
Inclusion Criteria:

* As above Either healthy or GI disease or non-GI disease

Exclusion Criteria:

* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: As above
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-11 (Estimated); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Construct validity measured by Validation of new score | 18 months
  Validation of new score

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Forbes, MD, Study Chair — UEA

IPD SHARING:
Plan to Share IPD: Undecided